CLINICAL TRIAL: NCT02013752
Title: Randomized Controlled Trial (RCT) of Primiparous Women Using the Modified Perineal Protection Device
Brief Title: The Effect of the Modified Perineal Protection Device During Delivery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Knut Haadem (Other)
Responsible Party: Sponsor-Investigator, Knut Haadem, M.D., PhD, Helsingborgs Hospital
Organization: Helsingborgs Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KH-HBG-13; ONLY-HBG (Registry Identifier: KH-HBG-13)
Record Dates: First submitted 2013-12-01; First posted 2013-12-17 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Perineal Tears.
Keywords: Delivery tears; Birth injuries; Perineal protection device
MeSH Terms: conditions — Birth Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perineal device during delivery (Active Comparator): Delivery should be managed by using the perineal protection device when the head was crowning and 5-6 cm of it was visible. One part the "tongue" was inserted between the head and the posterior vaginal wall and the "two wings" were held against the perineum and kept in place by the delivery attendant's hand.
  Interventions: Device: Perineal protection device.
- Standard care (Other): Standard care at delivery: Manual support of the perineum
  Interventions: Device: Perineal protection device.

INTERVENTIONS:
Device: Perineal protection device. — A device used to reduce perineal tears during delivery of the baby.
  Other Names: The perineal protection device have no brand name.

SUMMARY:
The purpose of this study is to determine whether a modified perineum protection device can reduce tearing during delivery.

DETAILED DESCRIPTION:
RCT investigation using a modified device during delivery of the baby's head (an earlier model has proved successful) and assess whether the use can decrease delivery tears as measured in length.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal delivery at term (week 36 - 41)

Exclusion Criteria:

* Age below 18
* Breech delivery
* Not understanding written and oral information

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Length of delivery tear measured in cm with ruler | at delivery - Participants will be followed for the duration of the first 24 hours
  The outcome measured is the occurrence of first and second degree vaginal and perineal tears during delivery.

SECONDARY OUTCOMES:
Adverse effects of the device on mother and child | at delivery-Participants will be followed for the duration of the first 24 hours
  Measure eventual adverse effects on mother and child.

CONTACTS AND LOCATIONS:
Overall Officials: Knut Haadem, M.D., PhD, Principal Investigator — Campus Helsingborg, Clinical Science Faculty of Medicine, Lund University, Helsingborg, Sweden
Locations (1):
- Dept Obstetrics and Gynecology, Helsingborg Hospital, Helsingborg, Skåne County, Sweden